CLINICAL TRIAL: NCT06745622
Title: A Multicenter, Open-label Study to Evaluate the Long-term Safety, Tolerability and Efficacy of HSK39297 in Patients With Paroxysmal Nocturnal Hemoglobinuria（PNH）
Brief Title: Long-term Safety and Tolerability of HSK39297 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK39297-203
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK39297 (Experimental)
  Interventions: Drug: HSK39297 tablets

INTERVENTIONS:
Drug: HSK39297 tablets — HSK39297 tablets until the end of treatment

SUMMARY:
This is a multicenter, open-label study to evaluate the long-term safety, tolerability and efficacy of HSK39297. Adult patients with PNH who had previously received and completed HSK39297 study treatment will be included. Eligible subjects can maintain HSK39297 treatment until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients With PNH who have previously received and completed HSK39297 treatment , and According to the researchers' judgment, the benefits of treatment outweigh the risks and may benefit from continued treatment with HSK39297;
2. Understand the study procedures and methods, voluntarily participate in this trial.

Exclusion Criteria:

1. Hereditary or acquired complement deficiency;
2. Active primary or secondary immunodeficiency;
3. History of splenectomy, bone marrow/ hematopoietic stem cell or solid organ transplants;
4. History of recurrent invasive infections caused by encapsulated organisms( e.g. meningococcus or pneumococcus) or Mycobacterium tuberculosis;
5. History of serious comorbidities that have been determined to be unsuitable for participation in the study;
6. Pregnant or Lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | through study completion，about 2 years

SECONDARY OUTCOMES:
Proportion of participants achieving hemoglobin levels ≥ 12 g/dL in the absence of red blood cell transfusions | through study completion，about 2 years
Change From Baseline in Hemoglobin in the absence of red blood cell transfusions | through study completion，about 2 years
Proportion of participants who remain free from transfusions | through study completion，about 2 years
Rate of breakthrough hemolysis (BTH) | through study completion，about 2 years
Proportion of participants with Major Adverse Vascular Events (MAVEs) | through study completion，about 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided